CLINICAL TRIAL: NCT05736900
Title: Counter-Regulatory Hormonal and Stress Systems in Patients With COVID-19
Acronym: CROSS-CO19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mingrone Geltrude, professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3223
Record Dates: First submitted 2023-02-20; First posted 2023-02-21 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with COVID-19 (Other): Patients admitted as in-patients with SARS-CoV-2 Infection
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — One samples of 5 mL blood is taken into a Serum tube for measurement of the RAAS-Biomarkers. After allowing to coagulate between 30 min and 60 min at room temperature, samples are centrifuged at 3000g for 10 min at room temperature.

SUMMARY:
The COVID-19 pandemic is associated with a highly variable presentation, ranging from patients who are asymptomatic or experience only mild symptoms to others with acute respiratory syndrome (ARDS) who require ventilatory support and carry a high risk of severe adverse outcomes and mortality. The most vulnerable population are older adults, usually people with chronic medical conditions and more often men than women.. Nevertheless, infection with SARS-CoV-2 can have deadly consequences even among those without any clear pre-existing medical conditions. Differences in adaptive immune responses and ensuing inflammatory reactions are proposed to contribute to the variable vulnerability to severe disease among patients infected with SARS-CoV-19. It is also possible that inter-individual differences in responsiveness of counter-regulatory hormonal and stress systems may further contribute to variable outcomes in infected patients, and that this may involve modulation of inflammatory responses. The hypothalamo-pituitary adrenal (HPA) axis in particular is a critical regulator of adaptive responses of metabolic and immune systems to various stressors, including. Sex-differences and age-related declines in adrenal cortical production of glucocorticoids and androgens as well as responsiveness of the HPA axis and immune function to stressors are particularly in older men. Such factors may contribute to the high morbidity associated with SARS-CoV-2 infection in elderly males.Among other important hormonal counter-regulatory systems, the renin angiotensin aldosterone system (RAAS) is prominently and directly impacted by SARS-CoV-2. Specifically both SARS-CoV-2 and SARS-CoV angiotensin-converting enzyme 2 (ACE2) to gain entry into cells. Tissue distrubtions of ACE2 match to viral distributions and systemic-wide impacts of SARS-CoV-2 or SARS-CoV beyond the lungs to kidneys, pancreas heart and other tissues. Studies in rats have shown that ACE2 is expressed in substantially higher amounts in alveolar epithelium, bronchiolar epithelium, endothelium and smooth muscle cells of pulmonary vessels of younger than older animals and among the latter group in higher amounts in females than males. Should the same apply to humans such differences may underly the predominance of symptomatic and more severe infections with both SARS-CoV-2 and SARS-CoV in older than younger patients, particularly male

DETAILED DESCRIPTION:
The evidence outlined above altogether favors the possibility that inbalance of the RAAS involving upregulated ACE and and angiotensin II and downregulated ACE2 and angiotensin 1-7 might be involved in the susceptibility of SARS-CoV-2 infected patients to more severe outcomes. Given links between the RAAS and the HPA axis with inflammatory processes [38-40], it is also possible that alterations in adrenal steroidal systems might further contribute to the highly variable responses to SARS-CoV-2 infection. This clinical protocol will therefore examine RAAS and the HPA stress system in SARS-CoV-2 infected patients with the objective of identifying differences in these counter-regulatory hormonal and stress systems that might explain progression to more severe disease in infected patients. With this and associated patient data (e.g., age, sex, comorbidities, medications) the plan is to also include application of artificial intelligence-based machine learning approaches to develop algorithms for prognostic prediction of disease outcomes. Given the forecasted numbers of deaths and secondary impacts on health even amongst those not infected, as well as the estimated more than one trillion dollar hit to the world economy, it is clearly important to identify effective treatments that may also be relevant to possible future outbreaks resistant to vacines developed based on the current pandemic. With this in mind the associated data should better facilitate identification of disease mechanisms that underly the more severe clinical phenotypes, thereby enabling educated identification of most appropriate therapeutic approaches for successful management of infected patients. Finally there is some evidence from the earlier SARS-CoV epidemic that infection with these coronaviruses may have health consequences well beyond the acute infection stage. By long-term follow-up, that also allows for inclusion of additional patients at follow-up, this protocol will further address concerns about chronic impacts on health among patients infected with the virus.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 years)
* Patients who meet on one or more of the following criteria for the screening test according to the CDC guidelines:
* Have fever or lower respiratory symptoms (cough, shortness of breath) and close contact with a confirmed COVID-19 case within the past 14 days; OR Have fever and lower respiratory symptoms (cough, shortness of breath) and a negative rapid flu test
* Patients with previous documented history of SARS-CoV-2 infection withn appropriate retrospectively collected andv available data.

Exclusion Criteria:

* Patients with impaired mental capacity that precludes informed consent
* Subjects who need medications that may interfere with or invalidate outcome parameters and that can not be stopped without significant risk (e.g., steroids, oral contraceptives)
* Severe or terminal co-morbidity which seriously interferes with possible treatment or health related quality of life
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
measure of the clinical status of patients at long-term follow up | 1 year
  This will be based on a composite cardiovascular and metabolic score that takes into account multiple clinical conditions known to be associated with SARS-CoV2 and SARS-CoV infections and hypothesized to be further worsened be infections. We will evaluate these scores using an established and widely implemented metabolic syndrome (MetS) severity Z-score (http://mets.health-outcomes-policy.ufl.edu). Clinical conditions will include diabetes mellitus, hypertension, ischemic heart disease, pulmonary disorders and any associated clinical complications that develop after infection (e.g., stroke, cardiac failure, death).

CONTACTS AND LOCATIONS:
Overall Officials: geltrude mingrone, Principal Investigator — Policlinico A. Gemelli IRCCS
Locations (1):
- Mingrone Geltrude, Roma, Italy

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Li G, Fan Y, Lai Y, Han T, Li Z, Zhou P, Pan P, Wang W, Hu D, Liu X, Zhang Q, Wu J. Coronavirus infections and immune responses. J Med Virol. 2020 Apr;92(4):424-432. doi: 10.1002/jmv.25685. Epub 2020 Feb 7. PMID 31981224
- [Background] Bornstein SR, Dalan R, Hopkins D, Mingrone G, Boehm BO. Endocrine and metabolic link to coronavirus infection. Nat Rev Endocrinol. 2020 Jun;16(6):297-298. doi: 10.1038/s41574-020-0353-9. PMID 32242089
- [Background] Sternberg EM, Chrousos GP, Wilder RL, Gold PW. The stress response and the regulation of inflammatory disease. Ann Intern Med. 1992 Nov 15;117(10):854-66. doi: 10.7326/0003-4819-117-10-854. PMID 1416562